CLINICAL TRIAL: NCT07189949
Title: A Phase I Study of HRS-2329 Evaluating Safety, Tolerability, and Pharmacokinetics in Subjects With Advanced Solid Tumors Harboring RAS Mutations or Amplifications
Brief Title: A Study of HRS-2329 in Participants With Advanced Solid Tumors Harboring RAS Mutations or Amplifications
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-2329-101
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors Harboring RAS Mutations or Amplifications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-2329 Group (Experimental)
  Interventions: Drug: HRS-2329 Tablet

INTERVENTIONS:
Drug: HRS-2329 Tablet — Oral HRS-2329 tablet.

SUMMARY:
This is an open-label, multi-center phase I clinical study to evaluate the safety, tolerability, and pharmacokinetics of HRS-2329 in participants with advanced solid tumors harboring RAS mutations or amplifications.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and are willing to sign the ICF, with good compliance and cooperation in follow-up;
2. Aged between 18-75 years old;
3. Participants with histologically/cytologically confirmed advanced solid tumors who have been previously tested or are confirmed by the central laboratory to harbor RAS mutations or amplifications and have failed standard treatment;
4. ECOG performance status (PS) score of 0 or 1;
5. Life expectancy > 3 months;
6. At least one measurable lesion per RECIST v1.1;
7. Adequate organ function.

Exclusion Criteria:

1. Toxicity (e.g., gastrointestinal reaction and skin toxicity) from prior anti-tumor treatment has not recovered to Grade ≤ 1 or a level specified in the inclusion/exclusion criteria;
2. Presence of central nervous system (CNS) metastases;
3. Participants with gastrointestinal diseases that affect drug administration/absorption;
4. Participants who have undergone major surgery other than diagnosis or biopsy within 28 days before the first dose, or are expected to undergo major surgery during the study period;
5. Presence of serious pulmonary diseases;
6. Active tuberculosis or a history of active tuberculosis infection within 48 weeks prior to screening, regardless of whether they have been treated;
7. Active or persistent gastrointestinal bleeding within 6 months prior to screening;
8. History of allogeneic bone marrow or solid organ transplantation;
9. History of deep vein thrombosis or pulmonary embolism within 6 months prior to screening;
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring clinical intervention;
11. Positive human immunodeficiency virus (HIV) (HIV1/2 antibodies), active chronic hepatitis B, or active hepatitis C (positive HCV antibody and positive HCV RNA);
12. Known history of hypersensitivity to any component of the drug product to be used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | From the screening period to 30 days after the last dose.
  Graded as per CTCAE v5.0.
Incidence and severity of serious adverse events (SAEs). | From the screening period to 30 days after the last dose.
  Graded as per CTCAE v5.0.
Dose-limiting toxicity (DLT). | From Day 1 to Day 21.
Maximum tolerated dose (MTD). | From Day 1 to Day 21.
Recommended Phase II Dose (RP2D). | 24 months.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax). | About 24 months.
The time to maximum concentration (Tmax). | About 24 months.
Area under concentration-time curve from time 0 to the last measurable concentration time point t (AUC0-t). | About 24 months.
Area under concentration-time curve from time 0 to infinity (AUC 0-∞). | About 24 months.
Apparent volume of distribution (Vz/F). | About 24 months.
Elimination half-life (t1/2). | About 24 months.
Apparent clearance (CL/F). | About 24 months.
Minimum concentration at steady state (Cmin, ss). | About 24 months.
Area under the blood concentration-time curve at steady state (AUCss). | About 24 months.
Accumulation ratio (Rac). | About 24 months.
Objective response rate (ORR). | About 24 months.
Duration of response (DoR). | About 24 months.
Disease control rate (DCR). | About 24 months.
Progression-free survival (PFS). | About 24 months.
Overall survival (OS). | About 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided